CLINICAL TRIAL: NCT02005263
Title: Hysteroscopic Assessment of Fallopian Tubal Patency
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Mississippi Medical Center (Other)
Responsible Party: Principal Investigator, John Preston Parry, MD, MPH, Assistant Professor, University of Mississippi Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2013-0230
Record Dates: First submitted 2013-12-03; First posted 2013-12-09 (Estimated); Last update posted 2017-11-08 (Actual); Status verified 2017-11

CONDITIONS: Infertility; Menorrhagia
Keywords: Hysteroscopy
MeSH Terms: conditions — Infertility; Menorrhagia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Salpingography (Experimental): Infusion of air bubbles through Fallopian tubes with hysteroscopic visualization; typically 1-2 mL is infused. This is less than that typically used in the established technique of sonosalpingography.
  Interventions: Procedure: Salpingography

INTERVENTIONS:
Procedure: Salpingography — Infusion of typically 1-2 mL of air bubbles in to the uterine cavity to assess whether they disappear through the ostia in to the Fallopian tubes.
  Other Names: Parryscope technique

SUMMARY:
Disease of the fallopian tubes is one of the most common reasons for infertility. The most common test, a hysterosalpingogram, tends to be painful,inconvenient, and frequently misses concurrent uterine disease. We propose using a less painful technique (through modified office hysteroscopy) for tubal assessment that can be performed in the office rather than hospital radiology and that uses gold standard technology for identifying coexisting uterine conditions.

ELIGIBILITY:
Inclusion Criteria:

1. 18 - 50 years old
2. Able to give consent
3. Must have a uterus
4. Must have documented negative testing for gonorrhea and chlamydia within the past year or previously negative when tested with a current partner in a monogamous relationship
5. Negative test prior to procedure

Exclusion Criteria:

1. Pregnancy
2. Active lower and upper genital tract infection
3. Patients with allergies to hysterosalpingogram contrast will not be exposed to a contrast material to which they are allergic
4. Premenarchal or postmenopausal
5. Unable to read English at a 6th grade level or above
6. History of endometrial Ablation
7. Asherman's syndrome > Stage 1

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 621 (Actual)
Dates: Start 2013-12; Primary Completion 2017-10-16 (Actual); Study Completion 2017-11-06 (Actual)

PRIMARY OUTCOMES:
Hysteroscopic assessment of tubal patency | 2 years
  Patients undergoing the procedure will be informed based on the findings as to whether or not it is believed that their Fallopian tubes are patent

CONTACTS AND LOCATIONS:
Overall Officials: John P. Parry, MD, Principal Investigator — University of Mississippi Medical Center
Locations (1):
- University of Mississippi Medical Center, Jackson, Mississippi, United States

REFERENCES:
- [Derived] Parry JP, Riche D, Rushing J, Linton B, Butler V, Lindheim SR. Performing the Parryscope technique gently for office tubal patency assessment. Fertil Steril. 2017 Oct;108(4):718. doi: 10.1016/j.fertnstert.2017.07.1159. Epub 2017 Aug 31. PMID 28843382